CLINICAL TRIAL: NCT07376798
Title: Effect of Patient Position on Bupivacaine Dose Requirement and Hemodynamic Stability in Spinal Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Balikesir Hospital Eduation and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: hduman
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Spinal Anesthesia; Hemodynamic Changes; Patient Positions; Bupivacaine
Keywords: Spinal Anesthesia; Bupivacaine; Patient Positioning; hemodynamic changes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor evaluating sensory block levels, motor block, and recording data will be blinded to group allocation. The anesthesiologist performing the spinal anesthesia and positioning cannot be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 8 mg Bupivacaine + Neutral Position (Active Comparator): Participants will receive 8 mg of 0.5% hyperbaric bupivacaine via spinal anesthesia at L3-4 or L4-5 interspace in sitting position. Immediately after injection, participants will be positioned supine in neutral (horizontal, 0°) position and maintained in this position throughout the procedure. Standard hemodynamic monitoring and management protocols will be applied.
  Interventions: Drug: Bupivacaine %0.5 (hyperbaric)
- 8 mg Bupivacaine + 10° Trendelenburg (Experimental): Participants will receive 8 mg of 0.5% hyperbaric bupivacaine via spinal anesthesia at L3-4 or L4-5 interspace in sitting position. Immediately after injection, participants will be positioned in 10° Trendelenburg position (head-down tilt) and maintained in this position throughout the procedure. Standard hemodynamic monitoring and management protocols will be applied.
  Interventions: Drug: Bupivacaine %0.5 (hyperbaric)
- 12 mg Bupivacaine + Neutral Position (Active Comparator): Participants will receive 12 mg of 0.5% hyperbaric bupivacaine via spinal anesthesia at L3-4 or L4-5 interspace in sitting position. Immediately after injection, participants will be positioned supine in neutral (horizontal, 0°) position and maintained in this position throughout the procedure. Standard hemodynamic monitoring and management protocols will be applied.
  Interventions: Drug: Bupivacaine %0.5 (hyperbaric)
- 12 mg Bupivacaine + 10° Trendelenburg (Experimental): Participants will receive 12 mg of 0.5% hyperbaric bupivacaine via spinal anesthesia at L3-4 or L4-5 interspace in sitting position. Immediately after injection, participants will be positioned in 10° Trendelenburg position (head-down tilt) and maintained in this position throughout the procedure. Standard hemodynamic monitoring and management protocols will be applied.
  Interventions: Drug: Bupivacaine %0.5 (hyperbaric)

INTERVENTIONS:
Drug: Bupivacaine %0.5 (hyperbaric) — 8 mg or 12 mg 0.5% hyperbaric bupivacaine administered intrathecally via spinal anesthesia at L3-4 or L4-5 interspace.

SUMMARY:
This study compares different combinations of local anesthetic doses and patient positions during spinal anesthesia for urogenital surgery. Spinal anesthesia is a common and safe technique where medication is injected into the lower back to numb the body during surgery.

The study will test two different doses of bupivacaine (a numbing medication): a lower dose (8 mg) and a standard dose (12 mg). It will also test two different patient positions after the spinal injection: lying flat (neutral position) and lying with the head slightly lower than the feet (Trendelenburg position).

Participants will be randomly assigned to one of four groups:

* Group 1: Lower dose + lying flat
* Group 2: Lower dose + head-down position
* Group 3: Standard dose + lying flat
* Group 4: Standard dose + head-down position

The study will measure how well the anesthesia works, how high the numbness spreads in the body, and how it affects blood pressure and heart rate. The goal is to find the best combination of dose and position that provides good anesthesia while keeping blood pressure stable.

This research may help doctors choose the safest and most effective anesthesia approach for each patient based on their individual needs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* American Society of Anesthesiologists (ASA) physical status classification I-II
* Scheduled for elective urogenital surgery
* Suitable candidate for spinal anesthesia
* Able to read, understand, and provide written informed consent
* Body Mass Index (BMI) less than 35 kg/m²
* Willing to participate in the study

Exclusion Criteria:

* Contraindications to spinal anesthesia (coagulopathy, infection at injection site, patient refusal)
* History of neurological disease
* Spinal deformity or previous spinal surgery
* History of allergic reaction to local anesthetics (amide-type)
* ASA physical status classification III or higher
* Emergency surgery
* Pregnancy
* Psychiatric illness preventing effective communication
* Refusal to participate in the study
* Unable to understand or provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Sensory Block Level | From injection to 30 minutes post-spinal anesthesia
  The highest dermatomal level of sensory blockade achieved, assessed using pin-prick test (sharp/dull discrimination). Measured as the specific dermatome level (e.g., T4, T6, T8).
Incidence of Hypotension | From spinal injection through end of surgery
  Proportion of participants experiencing hypotension, defined as mean arterial pressure (MAP) decrease ≥20% from baseline
Sensory Block Onset Time | From spinal injection through end of surgery
  Time required to achieve T10 dermatomal sensory block level, measured from completion of intrathecal injection to confirmation of T10 level by pin-prick test.

SECONDARY OUTCOMES:
Motor Block Degree | From spinal injection through end of surgery
  Degree of motor blockade assessed using modified Bromage scale (0=no motor block, able to raise extended leg; 1=unable to raise extended leg, able to flex knee; 2=unable to flex knee, able to flex ankle; 3=complete motor block, unable to move).
Surgical Adequacy | Throughout surgery
  Proportion of participants with adequate anesthesia for surgical procedure completion, assessed as adequate (surgery completed without supplemental analgesia/sedation) or inadequate (requiring supplemental intervention).
Incidence of Bradycardia | From spinal injection through end of surgery
  Proportion of participants experiencing bradycardia, defined as heart rate <50 beats per minute requiring treatment.
Incidence of Nausea and Vomiting | From spinal injection through end of surgery
  Proportion of participants experiencing nausea and/or vomiting during the intraoperative and immediate postoperative period.

IPD SHARING:
Plan to Share IPD: No